CLINICAL TRIAL: NCT03382548
Title: Reducing Antibiotics Treatment Duration for Ventilator-Associated Pneumonia
Brief Title: Defining Antibiotic Treatment Duration for Ventilator - Associated Lung Infection
Acronym: REGARD_VAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); Department for International Development, United Kingdom (Other Government); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAC17008
Record Dates: First submitted 2017-12-08; First posted 2017-12-26 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Ventilator Associated Pneumonia; Pneumonia, Bacterial
Keywords: Ventilator Associated Pneumonia; Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomisation will be done via stratified block randomisation by the study sites to ensure participants with similar characteristics such as gender and age are distributed equally in the intervention and control groups. Randomisation will be done with a computer programme with a seed to allow reproducibility. Randomisation will be done with a 1:1 ratio. To prevent predictability of the random sequence, generation of the randomisation sequence is performed by an independent statistician and details of the randomisation generation is unavailable to all investigators. Randomisation will be allocated using sequentially numbered opaque envelopes. Fitness criteria for randomisation must be met prior to randomisation.
Who Masked: Participant, Investigator
Masking Description: Patients will be blinded to the study, as they will not be informed of the treatment duration and likely to be sedated and unaware of the treatment regimens. Investigators will be blinded during the assessment of the participants for clinical stability based on the above-described criteria to minimise observer bias. Once conditions for stopping antibiotics are satisfied, the investigator will be unblinded and contact the primary physicians to stop antibiotics. The physicians will remain blinded until they are informed that the participant is suitable to stop antibiotics. Independent assessors, who are assigned to determine pneumonia recurrences, will be blinded from the randomisation arms. This will be achieved by blinding all study details, including randomisation arms, for participants with potential recurrences from these independent assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short antibiotic treatment duration for VAP (7 days or less) (Active Comparator)
  Interventions: Drug: Reducing Antibiotics treatment duration
- Long antibiotic treatment duration for VAP ( 8 days or more) (Active Comparator)
  Interventions: Drug: Standard Antibiotics treatment duration

INTERVENTIONS:
Drug: Reducing Antibiotics treatment duration — Antibiotics should be stopped from day 3 to 7 if respiratory cultures are negative and the patients fulfill a set of stringent clinical criteria signifying cardiopulmonary stability for 48 hours. If the respiratory cultures are positive, patients who fulfill the same set of clinical criteria should have their antibiotics stopped from day 5 to 7.
  Arms: Short antibiotic treatment duration for VAP (7 days or less)
Drug: Standard Antibiotics treatment duration — Participants in the control (long duration) arm will receive standard care, which is antibiotic treatment for at least 8 days with the exact duration decided by the primary physician.
  Arms: Long antibiotic treatment duration for VAP ( 8 days or more)

SUMMARY:
Intensive care units (ICUs), with high antibiotic consumption, are epicentres of antimicrobial resistance (AMR). Ventilator associated pneumonia (VAP) is the commonest hospital-acquired infection (HAI) in ICUs and is associated with a high morbidity and mortality in these vulnerable patients despite antibiotic therapy. No well-designed clinical trials studying antibiotic duration for VAP caused by predominantly non-fermenting Gram-negative bacteria have been conducted to date. Shortening antibiotic duration has the potential to improve individual patient outcomes and indirectly benefit other patients by reducing the selection pressure for multidrug resistant (MDR) bacteria within the ICU.

The study aims to demonstrate clinical non-inferiority-superiority of a short duration of antibiotics (up to 7 days) versus prolonged antibiotic therapy (as per physician preference) in adults with VAP in Asia. Patients who have been ventilated for more than 48 hours will be screened daily for signs and symptoms of VAP according to the US Centers for Disease Control and Prevention VAP criteria. Recruited patients will be reviewed daily for clinical signs of stability including temperature <38°C for 48 hours, systolic blood pressure >90mmHg without inotropes. Recruited patients will be randomised once they fulfill these clinical criteria of stability. In the intervention arm, antibiotics should be stopped within 7 days once the above criteria are fulfilled. In the control arm, antibiotics should be at least 7 days with the exact duration decided by the managing physicians.

The primary outcome of the study is a combined endpoint of mortality and VAP recurrence at day 60 of recruitment. The study hypothesis is that a shorter duration of treatment for VAP (7 days or less depending on clinical response) is not only noninferior, but may also be superior to a longer duration (8 days or more). The secondary outcomes of the study include clinical parameters such as rate of acquisition of MDRO hospital-acquired infections, duration of ventilation and hospitalization and days of antibiotics use. The study team will also characterise the microbiome changes in study participants according to the type and duration of antibiotics. MDROs collected will undergo whole genome sequencing for transmission dynamics study. The study is a multinational multicenter study involving hospitals in Asia.

Funder: The project will beis partly joinly funded by Medical Research Council/ Department for International Development (MRC/DfID) and Singapore National Medical Research Council (NMRC/CTG).

Grant Ref: MR/K006924/1 and MOH-000470 (MOH-CTGIIT18may-0003)

Conclusions This is a randomised controlled hierarchical non-inferiority-superiority trial being conducted in ICUs across Nepal, Thailand and Singapore. The primary outcome is a composite endpoint of death and pneumonia recurrence at day 60. Secondary outcomes include ventilator-associated events, multidrug-resistant organism infection or colonisation, total duration of antibiotic exposure, mechanical ventilation and hospitalisation. Adult patients who satisfy the US Centers for Disease Control and Prevention National Healthcare Safety Network VAP diagnostic criteria are enrolled. Participants are assessed daily until fever subsides for >48 hours and have stable blood pressure, then randomised to a short duration treatment strategy or a standard-of-care duration arm. Antibiotics may be stopped as early as day 3 if respiratory cultures are negative, and day 5 if respiratory cultures are positive in the short-course arm. Participants receiving standard-of-care will receive antibiotics for at least 8 days. Study participants are followed for 60 days after enrolment. An estimated 460 patients will be required to achieve 80% power to determine non-inferiority with a margin of 12%. All outcomes are compared by absolute risk differences. The conclusion of non-inferiority, and subsequently superiority, will be based on unadjusted and adjusted analyses in both the intention-to-treat and per-protocol populations.

Publication of this study

https://pubmed.ncbi.nlm.nih.gov/33986070/

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older
2. Invasive mechanical ventilation ≥ 48 hours
3. Satisfy the US Centers for Disease Control and Prevention National Healthcare Safety Network VAP diagnostic criteria

   * At least one of the following:

     1. temperature > 38 °C
     2. white blood cell count ≥ 12,000 cells/mm3 or ≤ 4,000 cells/mm3
     3. altered mental status with no other causes in >70 year-olds; AND
   * Two or more chest imaging tests demonstrating at least one of the following:

     1. new and progressive OR progressive and persistent infiltrate
     2. new and persistent OR progressive and persistent consolidation
     3. new and persistent OR progressive and persistent cavitation, AND
   * At least two of the following:

     1. new onset of purulent sputum, or change in character of sputum, or increased respiratory secretions, or increased in suctioning requirements
     2. new onset or worsening tachypnea or dyspnea
     3. rales or bronchial breath sounds
     4. worsening gas exchange defined by oxygen desaturations (e.g., PaO2/FiO2 <240), increased oxygen requirements or increased ventilation demand

Exclusion Criteria:

1. Poor likelihood of survival as defined by a Sepsis-related Organ Failure Assessment score (SOFA score) of >11 points
2. Immunocompromised patients (HIV with CD4 <200 cells/mm3, corticosteroids> 0.5 mg/kg per day for > 30 days, received chemotherapy in the past 3 months, solid organ or hematopoietic cell transplant)
3. Patients receiving antibiotic therapy for any other defined extra-pulmonary infections that warrant a duration of antibiotics longer than 7 days, or complications of pneumonia such as lung abscess or empyema, that warrant a duration of antibiotics longer than 7 days (excluding anti-tuberculosis treatment, antifungal medications, antibiotics meant for chronic suppression of chronic infections or chronic obstructive lung disease)
4. Patients who have been treated for VAP for more than 7 days from screening
5. Vulnerable population including prisoners and refugees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who suffered either death or pneumonia recurrence within 60(±5) days of enrolment | 60 days

SECONDARY OUTCOMES:
Proportion of patients who suffered ventilator-associated events within 60(±5) days of enrolment | 60 days
Duration of mechanical ventilation | 60 days
Duration of hospitalization | 60 days
Proportion of patients who acquired multidrug resistant infection or colonisation within 60(±5) days of enrolment | 60 days
Number of days of antibiotics during hospitalization | From 3 months before to 60 days after enrolment
Number and types of extrapulmonary infections during hospitalisation (determined from cultures taken from sterile sites) | 60 days
Characteristics of microbiota in terms of shifts in functional and metabolic capacity by comparing alpha and beta diversity metrics between the groups of patients | 3 years
Relative abundance of the genera in the microbiota between the groups of patients | 3 years
Route of transmission of MDR Gram-negatives in ICUs by comparing genomic sequencing data | 3 years
Quality Adjusted Life Years (QALY) loss | 3 years
  Mathematical modeling of antibiotic utilisation and sequencing data to predict outcomes
Financial costs | 3 years
  Mathematical modeling of antibiotic utilisation and sequencing data to predict outcomes

CONTACTS AND LOCATIONS:
Locations (7):
- Nepal (2):
  - Civil Hospital, Kathmandu
  - Patan Academy of Health Science, Patan Hospital, Kathmandu, Patan
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- Thailand (3):
  - Khon Kaen Hospital, Khon Kaen
  - Srinagarind Hospital, Khon Kaen
  - Sunpasitthiprasong Hospital, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: Yes
The clinical and laboratory data that are stored in our database may be shared with other researchers in the future. However, data will be anonymised and the researchers will not know your identity.

REFERENCES:
- [Derived] Mo Y, Booraphun S, Li AY, Domthong P, Kayastha G, Lau YH, Chetchotisakd P, Limmathurotsakul D, Tambyah PA, Cooper BS; REGARD-VAP investigators. Individualised, short-course antibiotic treatment versus usual long-course treatment for ventilator-associated pneumonia (REGARD-VAP): a multicentre, individually randomised, open-label, non-inferiority trial. Lancet Respir Med. 2024 May;12(5):399-408. doi: 10.1016/S2213-2600(23)00418-6. Epub 2024 Jan 22. PMID 38272050
- [Derived] Mo Y, West TE, MacLaren G, Booraphun S, Li AY, Kayastha G, Lau YH, Chew YT, Chetchotisakd P, Tambyah PA, Limmathurotsakul D, Cooper B. Reducing antibiotic treatment duration for ventilator-associated pneumonia (REGARD-VAP): a trial protocol for a randomised clinical trial. BMJ Open. 2021 May 13;11(5):e050105. doi: 10.1136/bmjopen-2021-050105. PMID 33986070
- See also: Mo Y, West TE, MacLaren G, et alReducing antibiotic treatment duration for ventilator-associated pneumonia (REGARD-VAP): a trial protocol for a randomised clinical trialBMJ Open 2021;11:e050105. doi: 10.1136/bmjopen-2021-050105 — https://bmjopen.bmj.com/content/11/5/e050105.citation-tools

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03382548/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03382548/SAP_003.pdf